CLINICAL TRIAL: NCT05749848
Title: Open-Label Study to Assess the Disposition of [14C]-LY3372689 Following Oral Administration in Healthy Male Participants
Brief Title: A Study of Carbon-14-Labelled [14C] LY3372689 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18430; I9X-MC-MTAF (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-02-20; First posted 2023-03-01 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Radiolabeled Drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [¹⁴C]-LY3372689 (Experimental): Single dose of [¹⁴C]-LY3372689 administered orally.
  Interventions: Drug: [¹⁴C]-LY3372689

INTERVENTIONS:
Drug: [¹⁴C]-LY3372689 — Administered orally.

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3372689), administered as a single dose that has the radioactive substance 14C incorporated into it, passes from blood into urine, feces and expired air in healthy male participants. The study will also measure how much of the study drug gets into the bloodstream, how its broken down, and how long it takes the body to get rid of it. The study will last about 4 weeks. Screening is required within 28 days prior to the start of the study and follow up is required approximately 7 days after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Male participants who are overtly healthy as determined by medical evaluation
* Have a body mass index within the range 18.5 to 32.0 kilograms per meter squared (kg/m²)
* Males who agree to use highly effective/effective methods of contraception for 14 weeks following the dose of LY3372689 may participate in this trial.

Exclusion Criteria:

* Have a clinically significant abnormal blood pressure and/or pulse rate as determined by the investigator at screening or check-in
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs
* Have evidence of significant active neuropsychiatric disease, as determined by the investigator
* Have participated in >3 radiolabeled drug studies in the last 12 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 8 (Actual)
Dates: Start 2023-02-24 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Urinary Excretion of LY3372689 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 17 post dose
  Urinary Excretion of LY3372689 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered
Fecal Excretion of LY3372689 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered | Predose up to Day 17 post dose
  Fecal Excretion of LY3372689 Radioactivity Over Time Expressed as a Percentage of the Total Radioactive Dose Administered

SECONDARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC (0-∞)) of Total Radioactivity and [¹⁴C]-LY3372689 | Predose up to Day 17 post dose
  PK: AUC (0-∞) of Total Radioactivity and [¹⁴C]-LY3372689
PK: Maximum Concentration (Cmax) of Total Radioactivity and [¹⁴C]-LY3372689 | Predose up to Day 17 post dose
  PK: Cmax of Total Radioactivity and [¹⁴C]-LY3372689
PK: Area Under the Concentration-Time Curve From Time Zero to Time (AUC (0-tlast)) of Total Radioactivity and [¹⁴C]-LY3372689 | Predose up to Day 17 post dose
  PK: AUC (0-tlast) of Total Radioactivity and [¹⁴C]-LY3372689
Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable) | Predose up to Day 17 post dose
  Total Radioactivity Recovered in Urine, Feces, and Expired Air (if applicable)
Total Number of Metabolites of LY3372689 | Predose up to 120 hour post dose
  Total Number of Metabolites of LY3372689

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- LabCorp CRU, Inc., Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No